CLINICAL TRIAL: NCT03557151
Title: Transdisciplinary Versus Usual Care for Type 1 Diabetes in Adolescence
Brief Title: Transdisciplinary Versus Usual Care for Type1 Diabetes in Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Melissa Alderfer, Principal Research Scientist and Associate Director, Center for Health Care Delivery Science, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DP3DK113235 (NIH); 1DP3DK113235-01 (NIH)
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: The study design randomizes participants to standard care or transdisciplinary care delivered through various modalities (in person; telehealth). Data collection occurs at 5 Time Points (0, 3, 6, 9 and 12 months).
Who Masked: Outcomes Assessor
Masking Description: Persons completing data scoring and entry tasks will be kept blinded to a given participant's treatment assignment. Most scoring is automated via the REDCap platform.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Usual Care participants will receive the same excellent multidisciplinary care they would receive at the same center were they not enrolled in the trial. In clinic visits scheduled at approximately 3-month intervals, they will see subspecialty board certified or eligible pediatric endocrinologists, supplemented as needed with involvement of certified diabetes educators, dietitians, social workers or psychologists. HbA1c target is < 7.5% with no severe hypoglycemia and acceptable quality of life. About half are expected to be on insulin pumps and carbohydrate counting, while the great majority of others are following basal-bolus multiple daily injection regimens, also based on carbohydrate counting. A rising proportion of patients use continuous glucose monitors and this trend is likely to accelerate during the study.
  Interventions: Other: Usual Care
- Transdisciplinary Care-In Person & Telehealth (Experimental): In addition to all elements of Usual Care, TC-IP participants will have follow-up clinic visits in-person or by telehealth at approximately 3 month intervals during the study that will consist of simultaneous involvement of an advanced practice nurse, dietitian and psychologist who will see the parent and adolescent together. TC team members will have passed a competency exam following completion of a training course on each of the TC team professional disciplines.
  Interventions: Behavioral: Transdisciplinary Care-In Person & Telehealth

INTERVENTIONS:
Other: Usual Care — Usual Care participants will receive the same excellent multidisciplinary Care they would receive at the same center were they not enrolled in the trial. In clinic visits scheduled at approximately 3-month intervals, they will see subspecialty board certified or eligible pediatric endocrinologists, supplemented as needed with involvement of certified diabetes educators, dietitians, social workers or psychologists. HbA1c target is < 7.5% with no severe hypoglycemia and acceptable quality of life. About half are expected to be on insulin pumps and carbohydrate counting, while the great majority of others are following basal-bolus multiple daily injection regimens, also based on carbohydrate counting. A rising proportion of patients use continuous glucose monitors and this trend is likely to accelerate during the study.
  Arms: Usual Care
Behavioral: Transdisciplinary Care-In Person & Telehealth — TC participants will receive all elements of the Usual Care intervention but they will do so in the context of face to face or telehealth delivery of TC follow-up visits with simultaneous involvement of an advanced practice nurse, dietitian and psychologist at each visit.
  Arms: Transdisciplinary Care-In Person & Telehealth

SUMMARY:
This study will consist of a randomized controlled trial to test a novel Transdisciplinary Care (TC) model of delivery of care for type 1 diabetes in adolescence. Adolescents and their parents/caregivers (n=150) will be randomized to Usual Care or TC care in a 1:2 ratio. Approximately half of those in TC care will received TC in person and half will receive it through telehealth. TC visits will consist of conjoint management of T1D by a TC team consisting of an Advanced Practice Nurse, Dietitian and Psychologist who will see parent-adolescent dyads together within the same visit. TC team members have trained each other in their respective disciplines. Outcome measures include glycohemoglobin (HbA1c) and questionnaires assessing diabetes self management behaviors. Other ancillary/exploratory measures are also completed.

DETAILED DESCRIPTION:
Large epidemiologic studies show that <25% of adolescents with type 1 diabetes (T1D) achieve targeted glycohemoglobin levels advocated by the American Diabetes Association (< 7.5%) or International Society of Pediatric and Adolescent Diabetes (< 7.0%). Optimal self-management of T1D requires daily insulin replacement by multiple injections or insulin pump, 4-6 daily blood glucose checks, regulation of carbohydrate intake and physical activity, prevention/correction of glycemic fluctuations and perhaps use of a continuous glucose monitor. This regimen places pervasive affective, behavioral, cognitive and social demands on adolescents with T1D and their families and psychosocial variables greatly impact their success in T1D self-care. Struggling with maintaining adequate glycemic control is essentially normative among adolescents, suggesting that conventional systems of care are not meeting the needs of this population. A substantial, growing literature provides an evidence base for psychosocial screening and behavioral intervention strategies targeting improved coping with the demands of T1D, but this evidence base has not penetrated fully into routine T1D care. Rigorous integration of this evidence into routine care for T1D could yield many benefits. Behavioral barriers to effective care are major concerns of all stakeholders, but conventional care is not well-equipped to address these issues. Concomitantly, the supply of board-certified pediatric endocrinologists is not keeping pace with growth of the T1D patient population, amplifying the need to validate alternative delivery systems that multiply the effective workforce of T1D health professionals. We will develop and test a novel Transdisciplinary Care (TC) approach (conjoint TC visits conducted by an Advanced Practice Nurse, Psychology Postdoctoral Fellow and Dietitian) to improve adolescents' T1D outcomes and justify a larger randomized controlled trial (RCT). In Year 1, crowdsourcing methods will engage youths with T1D, parents and health care providers (HCP) in planning a feasible, acceptable, safe and effective TC model that addresses youths' and families' psychosocial needs and capitalizes on the expertise of advanced practice nurses co-managing T1D with psychologists and dietitians. The Wallander et al. stress and coping model and the D'Zurilla and Goldfried problem solving model provide a sound conceptual framework for the TC model of care. The TC team will learn each discipline's skills in T1D management, develop a detailed TC manual to guide this work and others' future studies, see adolescents and parents together as a team, screen for potentially modifiable psychological impediments to T1D care, and promote families' coping resources by enhancing family-centered communication and problem solving, implementing empirically validated behavioral interventions and facilitating additional appropriate services for complex problems. Telehealth delivery of TC care carries several potential advantages, justifying its inclusion within a RCT comparing the effects of UC to TC delivered via various modalities on glycemic control and treatment adherence (primary outcomes) as well as quality of life and other psychosocial variables (exploratory outcomes). Qualitative and economic analyses will follow the RCT, providing perspectives on mechanisms of TC effects and its sustainability. Mixed qualitative and quantitative methods will validate an innovative model of T1D care for adolescents that could then be tested in a future definitive, multi-site RCT.

We will address these specific aims:

SPECIFIC AIM 1. In Year 1, with methods used effectively in our ongoing DP3 study of parents of children <6 years old with T1D, we will engage separate "crowds" of adolescents with T1D, parents, and HCPs in planning/refining a feasible, safe, acceptable and efficacious Trans-Disciplinary care model (TC) for T1D in adolescence. This crowdsourcing effort should yield a TC model that meets the needs of all key stakeholder groups, ensuring its feasibility, acceptance and efficacy.

SPECIFIC AIM 2. With study oversight by a diverse stakeholder panel and guided by a detailed intervention manual, 150 families of adolescents treated for T1D at Nemours practices in the Delaware Valley or Florida will participate in a rigorous Randomized Controlled Trial (RCT) in years 2 and 3. The RCT will compare Usual Care (UC) with Trans-Disciplinary Care on glycohemoglobin (HbA1C), treatment adherence, along with exploratory outcomes including health care use, T1D-related distress, quality of life, and treatment satisfaction. Delivery mode of Trans-Disciplinary Care will also be explored (e.g., Face-to-Face, Telehealth, Combined). The proposed trial will yield substantial information that could justify a definitive future test of this model, inform methodological planning for subsequent studies, and explore whether certain modes of delivery (e.g., Telehealth) are justified for evaluation in future trials.

SPECIFIC AIM 3. Qualitative interviews of adolescents, parents, and health care providers completed at the midpoint and end of the RCT will identify possible mediators or moderators of TC efficacy and guide refinements to the TC model. We will interview third party payers about the feasibility of dissemination of the TC model into practice and collect health care cost data. These analyses will strengthen the justification for a future, larger trial of TC, and guide refinements to the TC model to further enhance its efficacy.

ELIGIBILITY:
Adolescents:

* Age > 11 years but < 17 years at time of consent
* Diagnosis of Type 1 diabetes with duration of > 1 year
* Most recent HbA1C or mean HbA1C over the prior year 7.5-10.0%, inclusive
* Has had at least one clinic visit for T1D at a Nemours Children's Clinic within the past year
* Is not currently participating in any other research in which treatment adherence or glycemic control are study outcomes
* No T1D clinic visits in the preceding 12 months in which two or more care providers saw the patient together
* Is not on daily oral glucocorticoid treatment
* Is considered developmentally normal by the treating clinician (not in a self- contained special education classroom or been retained in 2 or more grades)
* Is able to read/comprehend study questionnaires in English
* Is not currently undergoing treatment for a coincident medical condition that, in the opinion of the treating physician, represents a contraindication to study participation
* Family must be able to access the internet

Parents:

* Is either a biological parent or legally appointed caregiver of the child
* Is the primary diabetes caregiver of the child: and at least weekly involvement in T1D care
* Routinely accompanies child for diabetes care at Nemours
* Is willing to schedule T1D clinic visits at a specific available location in Orlando or Wilmington
* Capable of participating in conversations in English during medical visits
* Anticipates continued medical care for T1D at Nemours for a year following study enrollment
* Is able to read/comprehend study questionnaires and decision aids in English
* Does not have an open abuse/neglect case with any child protection agency over the prior 3 years
* There is no evidence of frequent changes in the adolescent's household or living arrangements

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alderfer, PhD, Principal Investigator — Nemours Children's Clinic
Locations (3):
- United States (3):
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
A redacted data set stripped of all HIPAA-defined identifiers will be made available to interested and qualified researchers once all of the analyses of the study hypotheses have been completed and published. Access will require negotiation of a satisfactory Data Use Agreement between the Nemours Foundation and the interested party(ies).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Once analyses of primary study hypotheses have been completed and published, the de-identified data set will be available for 5 years.
Access Criteria: Contact the PI with a data use request and initiate a Data Use Agreement if the request is deemed to be feasible.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents with T1D and their caregiver were recruited and randomized as a dyad. 115 dyads (families) enrolled in the study
Pre-assignment Details: After enrollment, participants were required to complete baseline measures prior to randomization. A total of 11 families (22 participants) did not complete baseline measures and were not randomized to condition.
Groups:
- Usual Care: Usual Care includes the multidisciplinary health care, education and supports that are routinely available to Nemours families of youth with T1D. This includes clinic visits approximately every 3 months with a pediatric endocrinologist or advanced practice nurse, with referrals to a certified diabetes educator, dietitian, social worker or psychologist as deemed clinically necessary by that HCP.
- Transdisciplinary Care (In Person or Telehealth): Transdisciplinary Care includes all elements of Usual Care, but quarterly T1D visits are co-managed by an APN, RD and a Psychologist who provide care to the adolescent and parent(s) as a team during each visit. A central TC feature is active incorporation of evidence-based psychosocial care for T1D into visits including motivational interviewing techniques, systematic problem solving, and the facilitation of family communication to address each family's self-identified T1D challenges. TC visits will include interaction with all three team members jointly, with subsequent interaction between the parent/youth or both with a subset of this team as decided by family and team consensus during the visit.
Period: Randomization to 3 Months
Arm/Group | Usual Care | Transdisciplinary Care (In Person or Telehealth)
Started | 74 | 134
Adolescent Participants | 37 | 67
Caregiver Participants | 37 | 67
Completed | 72 | 132
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Period: 3 to 6 Months
Arm/Group | Usual Care | Transdisciplinary Care (In Person or Telehealth)
Started | 72 | 132
Adolescent Participants | 36 | 66
Caregiver Participants | 36 | 66
Completed | 72 | 132
Not Completed | 0 | 0
Period: 6 to 9 Months
Arm/Group | Usual Care | Transdisciplinary Care (In Person or Telehealth)
Started | 72 | 132
Adolescent Participants | 36 | 66
Caregiver Participants | 36 | 66
Completed | 70 | 132
Not Completed | 2 | 0
Not completed — moved out of state/discontinued care at Nemours | 2 | 0
Period: 9 to 12 Months (End of Study)
Arm/Group | Usual Care | Transdisciplinary Care (In Person or Telehealth)
Started | 70 | 132
Adolescent Participants | 35 | 66
Caregiver Participants | 35 | 66
Completed | 70 | 130
Not Completed | 0 | 2
Not completed — moved out of state/discontinued care at Nemours | 0 | 2

BASELINE CHARACTERISTICS:
Population: Adolescents with T1D and their caregivers were recruited and randomized to condition as a dyad. Diabetes-related medical variables (i.e., HbA1c) are only relevant for the adolescent participants and patient-reported outcomes (e.g., T1D treatment adherence, diabetes-related distress, diabetes-related quality of life) are reported separately by adolescents and caregivers and are reported here separately for these subsamples.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Transdisciplinary Care (In Person or Telehealth) | Total
Number analyzed (Participants) | 74 | 134 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Adolescents with T1D and their caregivers were recruited and randomized to condition as a dyad. Demographic information is being reported separately for participating adolescents and their caregivers. Two caregivers failed to report their age.
  years
    Adolescents: number analyzed (Participants) | 37 | 67 | 104
    Adolescents | 13.88 (1.77) | 14.07 (1.74) | 14.01 (1.75)
    Caregivers of adolescents: number analyzed (Participants) | 36 | 66 | 102
    Caregivers of adolescents | 42.61 (6.89) | 42.98 (7.06) | 42.85 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Adolescents with T1D and their caregivers were recruited and randomized as a dyad. Demographic information is being provided separately for adolescents and their caregivers. One caregiver did not provide their demographic information.
  Participants
    Adolescents: number analyzed (Participants) | 37 | 67 | 104
    Adolescents: Female | 19 | 36 | 55
    Adolescents: Male | 18 | 31 | 49
    Caregivers of adolescents: number analyzed (Participants) | 37 | 66 | 103
    Caregivers of adolescents: Female | 33 | 58 | 91
    Caregivers of adolescents: Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographic information is provided separately for adolescent participants and their caregivers.
  Participants
    Adolescents: number analyzed (Participants) | 37 | 67 | 104
    Adolescents: Hispanic or Latino | 8 | 11 | 19
    Adolescents: Not Hispanic or Latino | 29 | 54 | 83
    Adolescents: Unknown or Not Reported | 0 | 2 | 2
    Caregivers: number analyzed (Participants) | 37 | 67 | 104
    Caregivers: Hispanic or Latino | 6 | 11 | 17
    Caregivers: Not Hispanic or Latino | 31 | 55 | 86
    Caregivers: Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Adolescents with T1D and their caregivers were recruited and randomized as a dyad. Demographic information is presented separately for adolescent participants and their caregivers
  Participants
    Adolescents: number analyzed (Participants) | 37 | 67 | 104
    Adolescents: American Indian or Alaska Native | 0 | 0 | 0
    Adolescents: Asian | 1 | 0 | 1
    Adolescents: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adolescents: Black or African American | 5 | 13 | 18
    Adolescents: White | 23 | 43 | 66
    Adolescents: More than one race | 5 | 7 | 12
    Adolescents: Unknown or Not Reported | 3 | 4 | 7
    Caregivers of adolescents: number analyzed (Participants) | 37 | 67 | 104
    Caregivers of adolescents: American Indian or Alaska Native | 0 | 0 | 0
    Caregivers of adolescents: Asian | 0 | 0 | 0
    Caregivers of adolescents: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers of adolescents: Black or African American | 5 | 13 | 18
    Caregivers of adolescents: White | 26 | 43 | 69
    Caregivers of adolescents: More than one race | 1 | 6 | 7
    Caregivers of adolescents: Unknown or Not Reported | 5 | 5 | 10
HbA1c [Mean (Standard Deviation); unit: percentage glycosylated hemoglobin] — percentage glycosylated hemoglobin. Higher values indicate poorer glycemic control. Population: HbA1c was only collected for adolescent participants, not their caregivers
  percentage glycosylated hemoglobin
    number analyzed (Participants) | 37 | 67 | 104
    (all) | 8.52 (1.19) | 8.87 (1.26) | 8.74 (1.24)
Diabetes Self Management Profile - Youth Self Report [Mean (Standard Deviation); unit: score on a scale] — The Diabetes Self Management Profile - Self report version is completed by adolescents and assesses their adherence to T1D care. Total scores range from 0 to 84 points. Higher scores indicate better adherence/self-management Population: Two participants did not complete the measure at baseline
  score on a scale
    number analyzed (Participants) | 37 | 65 | 102
    (all) | 53.87 (12.33) | 52.37 (11.39) | 52.92 (11.70)
Diabetes Self Management Profile - Parent Proxy Report [Mean (Standard Deviation); unit: score on a scale] — The Diabetes Self Management Profile - Parent proxy version is completed by a caregiver and reports on their adolescent's adherence to T1D care. Total scores range from 0 to 84 points. Higher scores indicate better adherence. Population: This measure was completed by caregivers. One caregiver did not provide complete data on this measure at baseline
  score on a scale
    number analyzed (Participants) | 37 | 66 | 103
    (all) | 55.20 (12.1) | 53.68 (11.97) | 54.23 (11.98)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Hemoglobin (HbA1c)
Description: HbA1c expressed as percentage of glycosylated hemoglobin
Time Frame: baseline (enrollment; visit 1), 3 months (start of intervention; visit 2), 6 months (visit 3), 9 months (visit 4), 12 months (end of study; visit 5)
Population: These values are derived from blood work on the adolescent patients and represent all available raw data. HbA1c data were not available at all timepoints due to missed clinical visits and/or unreturned blood spot kits.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Usual Care | Transdisciplinary Care (In Person or Telehealth)
Number analyzed (Participants) | 37 | 67
percentage of glycosylated hemoglobin
  3 months: number analyzed (Participants) | 26 | 63
  3 months | 8.59 (1.56) | 9.02 (1.50)
  6 months: number analyzed (Participants) | 28 | 59
  6 months | 8.71 (1.41) | 9.03 (1.58)
  9 months: number analyzed (Participants) | 27 | 55
  9 months | 8.59 (1.66) | 8.98 (1.27)
  12 months: number analyzed (Participants) | 31 | 61
  12 months | 8.45 (1.21) | 8.97 (1.66)
Statistical Analysis 1: Comparison: Usual Care vs Transdisciplinary Care (In Person or Telehealth); Transdisciplinary Care is being compared to Usual Care using the Time 2 HbA1c (as baseline) and Time 5 HbA1c (as the outcome) controlling for race/ethnicity, gender, and age of the patient. The interaction of condition and time is used to evaluate the treatment effect. Missing data were not imputed; Test type: Superiority; p = 0.895, Mixed Models Analysis; Slope = -0.04, 95% CI 2-sided [-0.68 to 0.60], Standard Error of Mean 0.33

2. Secondary Outcome: Diabetes Self Management Profile-Self Report Form
Description: This 24 item measure assesses self-care behaviors that typify current T1D care. It is completed by the adolescent with T1D. Total scores are being used and range from 0 to 84 with higher scores indicating better adherence. In previous work, the scale had an internal consistency coefficient of .79 and a mean correlation of .48 with HbA1C.
Time Frame: baseline (enrollment; visit 1); 6 months (visit 3); 12 months (end of study, visit 5)
Population: These are raw data from all adolescent participants providing data. Decrements in the number of participants are due to missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Transdisciplinary Care (In Person or Telehealth)
Number analyzed (Participants) | 37 | 67
score on a scale
  6 month assessment: number analyzed (Participants) | 32 | 61
  6 month assessment | 53.45 (11.55) | 55.99 (11.86)
  12 month assessment: number analyzed (Participants) | 32 | 57
  12 month assessment | 53.97 (10.61) | 55.09 (12.09)
Statistical Analysis 1: Comparison: Usual Care vs Transdisciplinary Care (In Person or Telehealth); TC is being compared to UC using baseline and 12 month data, controlling for patient age, sex, and race/ethnicity. The interaction between condition and time is used to examine the treatment effect. Missing data were not imputed; Test type: Superiority; p = .33, Mixed Models Analysis; Slope = 2.29, 95% CI 2-sided [-2.29 to 6.88], Standard Error of Mean 2.34

3. Secondary Outcome: Diabetes Self Management Profile - Parent Proxy Report
Description: This 24 item parent-report measure parallels the youth self report measure and assesses self-care behaviors that typify current T1D care. The total scores is being reported with possible scores ranging from 0 to 84. Higher scores indicate better adherence to T1D care. In past work parent and youth reports have correlated at .63.
Time Frame: baseline (enrollment; visit 1); 6 months (visit 3); 12 months (end of study, visit 5)
Population: These are raw data. Discrepancies in participant numbers are due to missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Transdisciplinary Care (In Person or Telehealth)
Number analyzed (Participants) | 37 | 67
score on a scale
  6 month assessment: number analyzed (Participants) | 32 | 57
  6 month assessment | 53.73 (11.39) | 54.44 (12.27)
  12 month assessment: number analyzed (Participants) | 21 | 56
  12 month assessment | 52.67 (14.40) | 55.64 (13.72)
Statistical Analysis 1: Comparison: Usual Care vs Transdisciplinary Care (In Person or Telehealth); TC is being compared to UC using baseline and 12 month data and controlling for patient age, sex, and race/ethnicity. The interaction between condition and time is used to evaluate the treatment effect. Missing data are not imputed; Test type: Superiority; p = .07, Mixed Models Analysis; Slope = 4.1, 95% CI 2-sided [-.32 to 8.53], Standard Error of Mean 2.25

4. Other Pre Specified Outcome: Problem Areas in Diabetes (PAID) Scale - Adolescent Report
Description: This 14 item brief version of the scale measures problems, hassles, and distress related to diabetes and diabetes care. Respondents rate each item on a Likert-type scale ranging from 1 (not a problem) to 6 (serious problems). Scores range from 14 to 84 with higher scores indicating more diabetes-related problems.
Time Frame: Baseline (upon enrollment); 6 months; 12 months
Population: This adolescent-report measure was only completed by the adolescents taking part in the study (not caregivers). The data reported below are raw data (not imputed) and the discrepancies in the number of subjects are due to missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Usual Care: Usual Care participants receive the same excellent multidisciplinary care they would receive at the same center were they not enrolled in the trial. In clinic visits scheduled at approximately 3-month intervals, they will see subspecialty board certified or eligible pediatric endocrinologists, supplemented as needed with involvement of certified diabetes educators, dietitians, social workers or psychologists. HbA1c target is < 7.5% with no severe hypoglycemia and acceptable quality of life. About half are expected to be on insulin pumps and carbohydrate counting, while the great majority of others are following basal-bolus multiple daily injection regimens, also based on carbohydrate counting. A rising proportion of patients use continuous glucose monitors and this trend is likely to accelerate during the study.
Arm/Group | Usual Care | Transdisciplinary Care-In Person & Telehealth
Number analyzed (Participants) | 37 | 66
score on a scale
  Baseline | 38.73 (16.88) | 35.62 (16.45)
  6 months: number analyzed (Participants) | 33 | 63
  6 months | 39.57 (15.01) | 30.12 (13.97)
  12 months (end of study): number analyzed (Participants) | 32 | 59
  12 months (end of study) | 37.12 (17.16) | 30.55 (16.78)
Statistical Analysis 1: Comparison: Usual Care vs Transdisciplinary Care-In Person & Telehealth; This analysis included baseline and 12-month data. The interaction of condition (TC or UC) and time was used to examine the treatment effect. Child sex, age, and race/ethnicity were covariates. Missing data were not imputed; Test type: Superiority; p = .527, Mixed Models Analysis; Slope = -2.38, 95% CI 2-sided [-9.77 to 5.0], Standard Error of Mean 3.77

5. Other Pre Specified Outcome: Problem Areas in Diabetes (PAID) Scale - Caregiver Report
Description: This 15 item brief version of the scale measures problems, hassles, and distress related to diabetes and diabetes care. Respondents rate each item on a Likert-type scale ranging from 1 (not a problem) to 6 (serious problems). Scores range from 15 to 90 with higher scores indicating more diabetes-related problems.
Time Frame: Baseline (upon enrollment); 6 months; 12 months
Population: This caregiver-report measure was completed only by the caregiver participants in the study. Raw data are reported. Any deviations from the expected number of subjects is due to missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Transdisciplinary Care-In Person & Telehealth
Number analyzed (Participants) | 37 | 66
score on a scale
  Baseline | 52.85 (17.40) | 44.92 (19.73)
  6 months: number analyzed (Participants) | 33 | 62
  6 months | 54.42 (17.10) | 43.24 (19.44)
  12 months: number analyzed (Participants) | 33 | 60
  12 months | 53.46 (15.91) | 42.15 (18.16)
Statistical Analysis 1: Comparison: Usual Care vs Transdisciplinary Care-In Person & Telehealth; This analysis uses baseline and 12 month data. The interaction of condition and time is used to evaluate the treatment effect. Child sex, age, and race/ethnicity were used as covariates. Missing data were not imputed; Test type: Superiority; p = .253, Mixed Models Analysis; Slope = -3.30, 95% CI 2-sided [-8.94 to 2.35], Standard Error of Mean 2.89

6. Other Pre Specified Outcome: Type 1 Diabetes and Life (T1DAL) - Youth Self Report
Description: This measure assesses the adolescent's diabetes-related quality of life. Raw scores are converted to standardized scores that can range from 1 to 100. Higher scores indicate greater quality of life.
Time Frame: Baseline (upon enrollment); 6 months; 12 months (end of study)
Population: This youth-report measure was completed only by adolescent participants. Raw data are reported below. Any deviations in sample size are due to missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Transdisciplinary Care-In Person & Telehealth
Number analyzed (Participants) | 36 | 66
score on a scale
  Baseline | 61.84 (16.62) | 61.46 (18.21)
  6 months: number analyzed (Participants) | 31 | 62
  6 months | 57.85 (15.81) | 67.76 (18.74)
  12 months: number analyzed (Participants) | 30 | 58
  12 months | 57.76 (17.04) | 67.66 (19.71)
Statistical Analysis 1: Comparison: Usual Care vs Transdisciplinary Care-In Person & Telehealth; This analysis included baseline and 12 month data. The condition by time interaction was used to evaluate the treatment effect. Child age, sex, and race/ethnicity were included as covariates. Missing data were not imputed; Test type: Superiority; p = 0.01, Mixed Models Analysis; Slope = 9.69, 95% CI 2-sided [2.31 to 17.08], Standard Error of Mean 3.77

7. Other Pre Specified Outcome: Type 1 Diabetes and Life (T1DAL) Scale - Caregiver Report
Description: This caregiver-report measure assesses caregiver quality of life related to their child's diabetes. Raw scores are standardized to range from 0 to 100 with higher scores indicating better quality of life.
Time Frame: Baseline (upon enrollment); 6 months; 12 months (end of study)
Population: This caregiver-report measure was only completed by caregiver participants. Raw data is presented. Any deviations in the number of subjects across time points is due to missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Transdisciplinary Care-In Person & Telehealth
Number analyzed (Participants) | 37 | 66
score on a scale
  Baseline | 55.97 (11.50) | 65.64 (14.74)
  6 months: number analyzed (Participants) | 33 | 60
  6 months | 56.62 (10.10) | 66.73 (14.54)
  12 months: number analyzed (Participants) | 33 | 56
  12 months | 55.36 (11.20) | 66.32 (15.80)
Statistical Analysis 1: Comparison: Usual Care vs Transdisciplinary Care-In Person & Telehealth; This analysis uses baseline and 12-month data. The interaction between condition and time is used to evaluate the treatment effect. Child age, sex, and race/ethnicity were covariates. Missing data were not imputed; Test type: Superiority; p = .83, Mixed Models Analysis; Slope = .45, 95% CI 2-sided [-3.62 to 4.35], Standard Error of Mean 2.07

ADVERSE EVENTS:
Time Frame: Approximately 1 year. Adverse events (AEs) were recorded for adolescent participants from the time of randomization through final study visit or close of final study visit time window. AEs were not collected regarding caregivers. Of note, the report of AEs for those randomized to Transdisciplinary Care (TC) includes the 3 month time period AFTER randomization but PRIOR to receiving the intervention. It also includes 6 participants who were randomized to but never attended a TC visit.
Description: ClinicalTrials.gov definitions are being used. Serious Adverse Events include hospitalizations for any reason and emergency room visits related to diabetes care.
Arm/Group | Usual Care | Transdisciplinary Care (In Person or Telehealth)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/67
Serious Adverse Events (participants affected / at risk) | 3/37 | 7/67
Other Adverse Events (participants affected / at risk) | 18/37 | 26/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=37) | Transdisciplinary Care (In Person or Telehealth) (N=67)
Inpatient Hospitalization related to diabetes (Endocrine disorders) | 1 (1) | 3 (3) — Two instances of the AE reported for those randomized to TC occurred prior to beginning the intervention (1 patient) or after opting out of TC and returning to Usual Care (1 patient)
Emergency Room visit related to diabetes (Endocrine disorders) | 1 (1) | 6 (8) — One instance of this AE occurred for a patient randomized to TC before receiving the intervention. Two additional instances of this AE occurred for a patient randomized to TC who opted to return to Usual Care prior to receiving any TC care visits
Inpatient Hospitalization unrelated to diabetes (General disorders) | 1 (1) | 1 (1) — Instances included appendicitis and injury
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=37) | Transdisciplinary Care (In Person or Telehealth) (N=67)
Increase of 1.5% or more in HbA1c from one data point to another during study participation (Endocrine disorders) | 7 (14) | 19 (28) — Seven instances of this AE were reported among 7 TC participants prior to their receipt of the TC intervention. Two additionally instances occurred among 2 participants randomized to TC but opting to return to Usual Care prior to receiving TC
Decrease in QoL of 1.5SD or more (General disorders) | 8 (8) | 7 (8) — Two instances of this AE (drop from baseline to 6 months and drop from baseline to 12 months) were reported by 1 participant randomized to TC but who opted to return to Usual Care before receiving TC
Gap in clinical care of 6 months or more (Surgical and medical procedures) | 8 (9) | 5 (5) — All instances of this AE reported for participants randomized to TC occurred after the participant opted out of the assigned intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03557151/Prot_SAP_001.pdf